CLINICAL TRIAL: NCT06212180
Title: Comparison of the Comfort of Patients Under Non-invasive Ventilation According to the Use of a Sub Nasal Mask Versus an Oronasal Mask
Brief Title: Comfort of Patients Under Non Invasive Ventilation According to the Mask
Acronym: ComPaNIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231673; 2023-A02093-42 (Other: ID-RCB)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: COPD Exacerbation; Hypercapnia; Hypoventilation Obesity Syndrome; Acute Respiratory Failure
Keywords: Non-invasive ventilation; Acute respiratory failure; Comfort
MeSH Terms: conditions — Hypercapnia; Obesity Hypoventilation Syndrome | interventions — Masks

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mask — patients will be their own comparator. Patients will try both mask for 10 min and then decide which mask they want for the rest of the ventilation
  Other Names: oronasal mask or subnasal mask

SUMMARY:
A sub-nasal mask with a skirt that fits the nostrils and with a dedicated port for the nasogastric tube has recently been introduced. This interface has never been compared to nasal-oral masks. We hypothesise that such a sub-nasal mask increases comfort compared to a conventional naso-oral mask. The primary objective is to compare the comfort of the sub-nasal mask with that of a standard naso-oral mask.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is a first-line treatment for many conditions encountered in the ICU. This technique requires training of heath professionals, appropriate equipment, optimisation of ventilator settings and good cooperation from the patient. Indeed, NIV failures lead ton invasive mechanical ventilation, thus increasing morbidity and mortality. These failures are favoured by the patient's poor tolerance to NIV. The success of the treatment depends greatly on the patient's compliance and comfort. The choice of the mask is therefore essential. There are different types of interface, such as the full-face helmet, the face mask, the nasal-oral mask or the nasal mask. The nasal-oral mask rmains the most commonly used interface. Recommendations emphasise the importance of choosing a mask that is the right size and best tolerated by the patient. Despite benefits of NIV, there are a number of potential complications: skin lesions at pressure points, particulaly at the nasal bridge, gastric distension, barotrauma, haemodynamic effects of positive presure ventilation, claustrophobia, anxiety, difficulty in speaking and eating, dry eyes, patient-ventilator asynchrony. Some of these complications depend on the type of mask used. a sub-nasal mask with a skirt that fits the nostrils and a dedicated port for the nasogastric tube has recently been introduced. To our knowledge, this interface has never been compared to commercially avaible nasal-oral masks.

ELIGIBILITY:
Inclusion Criteria:

Indication of NIV, carried out by the physicians in charge of the patient, among the following:

* COPD exacerbation
* Hydrostatic acute pulmonary edema
* Acute Chest Syndrome with Hypercapnia in Sickle Cell Patients
* Post-extubation, planned in a patient at risk or recovering from extubation failure
* Hypoventilation-obesity syndrome

Exclusion Criteria:

Formal contraindication to NIV among:

* Indication for orotracheal intubation at the outset
* Non-cooperative, agitated, opponent of the technique
* Coma
* Respiratory exhaustion
* Shock, severe ventricular arrhythmias, immediate aftermath of cardiac arrest
* Undrained pneumothorax, blowing chest wound
* Upper airway obstruction (except sleep apnea, laryngotracheomalacia)
* Uncontrollable vomiting
* Upper gastrointestinal bleeding
* Measure of protection of justice
* Facial deformity
* Dying or palliative care patient
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in intensive care, continuous monitoring unit or pulmonary intensive care with an indication for NIV.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
1 to 10 self assessment scale | throughout the study (an average of 10 months)
  Comfort will be assessed by a numerical self-assessment scale from 0 to 10.

SECONDARY OUTCOMES:
Percentage of subjects who prefer one type of mask over the other | throughout the study (an average of 10 months)
Percentage of leakage volume compared to the tidal leakage volume | throughout the study (an average of 10 months)
Dyspnea | throughout the study (an average of 10 months)
Number of interventions on mask position by nurses during NIV session | throughout the study (an average of 10 months)
Number of side effects | throughout the study (an average of 10 months)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CARPENTIER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, Hôpital Bicêtre
Locations (3):
- France (3):
  - Hôpital Henri Mondor - Réanimation/ Unité de Surveillance Continue, Créteil
  - CHU Bicêtre - Unité de Soins Intensifs Pneumologique, Le Kremlin-Bicêtre
  - CHU Bicêtre - USC, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: No